CLINICAL TRIAL: NCT06371742
Title: The Effect of Fluid Intake on the Duration of Labour, Type of Delivery, Well-being of the Pregnant Woman and the Newborn
Brief Title: Study of the Fluid Intake Effect During Labour
Status: Completed | Type: Observational
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Other Study IDs: 539HydrationNutr
Record Dates: First submitted 2024-03-27; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Labor Complication
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Liquid ingestion during labour — An assessment of the volume capacity of the water glasses was carried out using duly certified 50mL syringes in order to calibrate and control the correct measurement of the amount of water ingested. Water is measured using a graduated cup, which is pre-existing in the BP service, since its water intake policy is governed by the formula 1ml/kg/h of clear liquids (water or tea).

SUMMARY:
Ingestion during labor is an issue that has attracted the attention of the scientific community in recent decades, with different practices occurring in different countries. However, the scientific evidence of the risk / benefit of fluid intake in labor is still not fully understood. The aim of this study was to contribute with data that allow the evaluation of an eventual relationship between the amount of fluid ingested during labor and the type of delivery, the duration of labor, the occurrence of nausea and vomiting and the value of the Index of Apgar at the 1st and 5th minutes of the newborn's life. An observational study, with a convenience sample of 144 parturient from two hospitals of Portugal were employed. The analysis was based on recording the before mentioned variables and potentially confounding variables. In order to control for potential sources of bias in the study and to guarantee the homogeneity of the sample in the specific statistical treatment of each dependent variable, an observation grid was drawn up for all the participants in the study. Twenty eight of the parturient, the parturient's ambulation, labour analgesia, food intake during labour, the use of oxytocin during labour, the occurrence of postpartum complications, the birth weight of the newborn and the occurrence of birth complications.

DETAILED DESCRIPTION:
To carry out the study, authorization was requested from the National Data Protection Commission. Each participant was given a code to ensure the confidentiality and protection of the data collected. The data obtained was recorded on coded sheets (without any element identifying the participant) and entered into a database accessed only by the researcher in charge and processed using the identification code assigned to the participants. The study was also authorized by the Ethics Committee of the Egas Moniz School of Health and Science, by the Ethics Committee of Garcia de Orta Hospital, and by Barreiro Hospital. The data was collected after the informed consent of the pregnant woman/couple, using an observation grid that allowed the variables to be observed and recorded, in accordance with the Declaration of Helsinki.

This is an observational study, since the researcher chose not to interfere in the clinical practice of each of the hospital institutions, and nothing was imposed on the pregnant woman/couple.

The analysis was based on recording the variables mentioned above and potentially confounding variables. In order to control for potential sources of bias in the study and to guarantee the homogeneity of the sample in the specific statistical treatment of each dependent variable, an observation grid was drawn up for all the participants in the study, including, in addition to the amount and type of fluid ingested, the type of labour, the assessment of the duration of labour, expressed in the partogram (a sheet recording the progress of labour) in the parturient's file, the occurrence of nausea and vomiting during labour. Apguar index (AI) at the first and fifth minute of life, the age of the parturient, the parturient's ambulation, labour analgesia, food intake during labour, the use of oxytocin during labour, the occurrence of complications in the postpartum period, the weight of the Newborn (NB) at birth and the occurrence of complications during labour.

The target population was primiparous women with low-risk, full-term pregnancies with cephalic fetuses and spontaneous onset of labour. The sample size was determined by the Gpower 3.1® programme, according to the statistical analysis to be carried out and with a 95% confidence interval, which suggested an sample number of 150. This was a convenience sample made up of pregnant women who had signed an informed consent form at Garcia de Orta Hospital and at Barreiro Hospital and who met the inclusion criteria. All parturients with associated pathologies, either previous or during pregnancy, medium or high-risk pregnancies and who develop problems during labour, such as hyperthermia, hypotension, hypoglycaemia, lipothymia, fetuses with cardiotocographic alterations and NB with tight cervical circles at birth were excluded. Pregnant women who did not walk and who were not given intravenous oxytocin during labour were also excluded in order to standardize the sample, as were all the parturients who did not consent to their data being used.

An assessment was made of the volume capacity of the water glasses, using duly certified 50 mL syringes, in order to calibrate and control the correct measurement of the amount of water ingested. The water was measured using a graduated glass, since its water intake policy is governed by the formula 1ml/kg/hour of clear liquids (water or tea). Subsequently, an observation grid was drawn up for all the participants in the study, and the data was collected and integrated into the observation grid directly from the pregnant women present in the delivery room.

The data was processed and analysed statistically using IBM SPSS™ version 24 software. Taking into account the data collected on the observation grid, the sample was descriptively analysed, the assumptions for applying statistical methods were checked and the data was statistically analysed. Bearing in mind the objectives of this study [to see if there is an association between the amount of water ingested during labour (LW) and the type of delivery, the duration of LW, the occurrence of nausea and vomiting, the Apgar score (AI) at the 1st and 5th minute of life of the Newborn (NB)] and the different nature of the variables: scalar - total amount of fluid ingested (mL), duration of labour (hours) and nominal - type of delivery; occurrence of nausea and vomiting; AI at the 1st and 5th minutes, different statistical analyses were used to confirm the null hypothesis as well as testing the normality of the sample distribution for the scalar variables (duration of labour) using the Kolmogorov-Smirnov and Shapiro-Wilk tests. As the distribution of the variable was not normal ρ ≤ 0.05. The investigators analysed it using non-parametric tests using Spearman's Rho Correlation Coefficient. For the remaining variables, the Logistic Regression test was applied, since this statistical analysis makes it possible to estimate the chances of a given event occurring, given a set of variables. In this case, for example, to identify the risk of dystocia for each mL of fluid ingested.

ELIGIBILITY:
Inclusion Criteria:

* low-risk pregnancies
* term pregnancies (> 37 weeks gestation),
* primiparous pregnancies
* fetuses with cephalic presentation
* with spontaneous onset of labour
* at the beginning of the active phase of labour (> 4cm dilation).

Exclusion Criteria:

* parturients with associated pathologies, either previous or during pregnancy, medium or high-risk pregnancies and who develop problems during labour, such as hyperthermia, hypothermia, hypoglycaemia, lipothymia, foetuses with cardiotocographic alterations and NBs with tight cervical circles at birth.
* pregnant women who did not walk and who were not given intravenous (IV) oxytocin during labour
* parturients who did not consent to their data being used.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: An initial analysis of the data collected from the total sample of N=171 showed that 16 per cent (N=27) of parturients did not walk (N=10) or were not given oxytocin (N=17). The use of ambulation and oxytocin speeds up the labour process. Therefore, in order to control labour conditions and external influences, as well as to guarantee the homogeneity of the sample, pregnant women who did not walk or were not given oxytocin were excluded. Therefore, the overall sample considered for the descriptive analysis was N= 144.
  The overall sample was made up of pregnant women aged between 18 (10.4%) and 39 (0.7%), with an average age of 26.22 ± 5.42. The average weight of the pregnant women was 74.06kg ± 11.62, ranging from 52 (1.4%) to 122kg (0.7%), with the average being 70kg (7.6%).
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Type of labour | During the labour
  The labour type was registered taken in account if eutocic, cup, forceps, caesarean section.
Duration of labour | During the labour
  The mean value of labour duration in hours (h)
Occurrence of nausea and vomiting | During the labour
  The frequency of nausea and vomiting episodes in number
Apgar index of the newborn (From 0 to 10) | At the 1st and 5th minute of the newborn's life
  The apgar index will be analysed by a score from 0 to 10. The 5-minute Apgar score of 7-10 as reassuring, a score of 4-6 as moderately abnormal, and a score of 0-3 as low in the term infant and late-preterm infant and as a nonspecific sign of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Bernardo, PhD, Principal Investigator — Egas Moniz School of Health and Science
Locations (1):
- Egas Moniz School of Health and Science, Almada, Monte de Caparica, Portugal